CLINICAL TRIAL: NCT04643015
Title: New Image Techniques for Magnetic Resonance Imaging in Children and Adults
Brief Title: New Ways of Doing Magnetic Resonance Imaging in Children and Adults
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 20-482
Record Dates: First submitted 2020-11-19; First posted 2020-11-24 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Pediatric Disorder; Adult Disease
Keywords: Magnetic Resonance Imaging; MRI; 20-482; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Participants: Patients of any age, including males and females, who are being treated in the Department of Pediatrics and are already scheduled to undergo MRI
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — Briefly, new MRI sequences will be used on a patient who is undergoing a scheduled, clinically necessary MRI exam. Any new research sequence will be scanned in addition to the clinically required sequences and will not interfere with the clinical scan other than requiring five to ten minutes of additional "table time". There will be no invasive measures under this protocol.

SUMMARY:
This study is being done to see how we can prevent problems caused by movement during the MRI scan. Different ways of doing the scan (techniques) will be tested to see if they are practical and can prevent problems related to motion. For example, changes in the timing of the magnetic field and the radio waves will be examined, and at changes in the way a computer is used to process the images. The new techniques will be compared with the techniques that are usually used.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any age, including males and females, who are being treated in the Department of Pediatrics and are already scheduled to undergo MRI

Exclusion Criteria:

* Anyone who would normally be excluded from undergoing an MRI examination as per Memorial Hospital for Cancer and Allied Diseases Screening Questionnaire for MRI (Appendix A). Subjects with pacemakers or aneurysm clips that are MRI conditional or MRI compatible may enroll in the study if the study is clinically indicated.
* Female patients who are pregnant
* Patients who are unable to comply or complete the MRI exam due to claustrophobia or high levels of anxiety
* Patients at higher risk due to age, frailty, or the emergent nature of their condition
* Patients who are undergoing MRI only of the head, neck or spine

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Potential research subjects will be identified by a member of the patient's treatment team, the protocol investigator, or research team at Memorial Sloan-Kettering Cancer Center (MSK). With consultation of the clinical team, the investigator or a consenting professional from the research team will go to the treating physician's clinic to discuss the study and consent the patient in person.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2026-11-18 (Estimated); Study Completion 2026-11-18 (Estimated)

PRIMARY OUTCOMES:
Compare Image Quality | Day of MRI
  To assess the new MRI sequences or MRI analysis methods and compare their image quality to current clinical ones. Specifically, we aim to compare the routine sequences with the experimental sequences.

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Behr, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

DOCUMENTS (1):
  • Informed Consent Form (2022-02-08): https://cdn.clinicaltrials.gov/large-docs/15/NCT04643015/ICF_000.pdf